CLINICAL TRIAL: NCT02891109
Title: The Role of Regulatory B Cells in the Chronic Immune Thrombocytopenia
Brief Title: Regulatory B Cells and Chronic Immune Thrombocytopenia
Acronym: PTIREG
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PTIREG
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic; Regulatory B Cells
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients group: Adults patients with chronic immune thrombocytopenia
  Interventions: Biological: Biological tests
- control group: Adults without immune thrombocytopenia
  Interventions: Biological: Biological tests

INTERVENTIONS:
Biological: Biological tests — From the blood: B and T cells extraction then co-culture B and T cells and characterization of lymphocytes by flow cytometry

SUMMARY:
The chronic immune thrombopenia is an autoimmune disease caused by B cells. These cells produce anti platelets and megakaryocytes antibodies. Some B cells, named regulatory B cells, are known to control other cells. Their action in chronic immune thrombopenia is actually unknown.

DETAILED DESCRIPTION:
The chronic immune thrombopenia is an autoimmune disease caused by B cells. These cells produce anti platelets and megakaryocytes antibodies. Some B cells, named regulatory B cells, are known to control other cells. Their action in chronic immune thrombopenia is actually unknown. In our cohort of chronic immune thrombopenia and controls, we realized a flow cytometry analyze of B and T cells and a co-culture to determine regulatory B cells functionality.

ELIGIBILITY:
Inclusion Criteria:

* Purpura, Thrombocytopenic, Idiopathic, chronic phase (>12 months)
* no treatment or thrombopoietin receptor agonists

Exclusion Criteria:

* < 18 years
* Purpura, Thrombocytopenic, Idiopathic, acute phase
* pregnancy
* others causes of thrombopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with a Purpura, Thrombocytopenic, Idiopathic, in chronic phase (>12 months) and healthy volunteers as control residents in Brest town, France.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Regulatory B cells functionality | 1 week
  inhibition of T cells proliferation with co-culture B and T cells

SECONDARY OUTCOMES:
Cytometry immunophenotyping of B and T cells | 1 week
  characterization of B and T cells by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Jamin, PhD, Principal Investigator — CHRU de Brest; Lenaig Le Clech, MD, Principal Investigator — CHRU Brest; Brigitte Pan-Petesh, MD, Principal Investigator — CHRU Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No